CLINICAL TRIAL: NCT05110339
Title: Efficacy of Dexmedetomidine on Postoperative Analgesia After Radical Mastectomy: Randomized Controlled Trial
Brief Title: Efficacy of Dexmedetomidine on Postoperative Analgesia
Acronym: EDPARMRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Tamaulipas (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCAECV01
Record Dates: First submitted 2021-10-12; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: A prospective randomized double-blinded study
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessor did not know the allocation of the participants. The patient is not informed of the medication used in the erector spinae block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine plus Dexmedetomidine (Experimental): In addition to standard general anesthesia, patients receive erector spinae block with ropivacaine at a dose of 0.5% plus dexmedetomidine at 0.3 mcg / kg corrected in a volume of 20 ml at the level of thoracic vertebra number 4, guided with ultrasound and under sterile technique, the date and time of application are recorded on the data collection sheet.
  Interventions: Drug: Ropivacaine plus dexmedetomidine
- Control group (Active Comparator): In addition to standard general anesthesia, patients receive erector spinae block with ropivacaine at a dose of 0.5% in a volume of 20 ml at the level of thoracic vertebra number 4, guided with ultrasound and under sterile technique, the date and time of application are recorded on the data collection sheet.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine plus dexmedetomidine — Erector spinae block with ropivacaine at a dose of 0.5% plus dexmedetomidine at 0.3 mcg / kg.
  Arms: Ropivacaine plus Dexmedetomidine
Drug: Ropivacaine — Erector spinae block with ropivacaine at a dose of 0.5%.
  Arms: Control group

SUMMARY:
This prospective, randomized, double-blind study is designed to evaluate the postoperative analgesic efficacy of dexmedetomidine as an adjunct to ropivacaine in erector spinae block in patients undergoing radical mastectomy. The investigators hypothesis is that the administration of ropivacaine 0.5% associated with dexmedetomidine in the blockade via the plane in the erector spinae is less effective in controlling acute postoperative pain in radical mastectomy than the administration of ropivacaine 0.5% without dexmedetomidine.

DETAILED DESCRIPTION:
Patients undergoing radical mastectomy are randomly assigned to receive, in addition to standard general anesthesia, a block of the erector spinae plane with ropivacaine at a dose of 0.5% for the control group (n = 13) and ropivacaine at a dose of 0.5% more dexmedetomidine at 0.3 mcg kg (n = 15) for the intervention group. General anesthesia was induced using anxiolysis with midazolam at 30 mcg / kg corrected weight, as induction, propofol at a dose of 1.5 - 2 mg kg, opioid analgesia with fentanyl at a dose of 3 mcg / kg weight corrected with 30% according to ideal weight initial bolus dose, and dose as required, neuromuscular relaxation with cisatracurium at a dose of 0.1 mg / kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radical mastectomy for pathology "breast cancer"
* Patient undergoing anesthetic technique due to erector spinae plane block
* Informed consent to perform the anesthesia technique.
* Karnofsky> 80 points

Exclusion Criteria:

* Emergency surgery
* Patient with mental pathology that prevents pain assessment.
* Rejection of anesthetic technique.
* Patient with allergy to local anesthetics
* Patient with local infection of the puncture site for application of the erector spinae block

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain score | 0 hours
  The intensity of pain is evaluated by the visual analog scale (VAS) that measures pain severity expressed on a numerical scale of 0-10: 0, "no pain"; 10, "worst pain imaginable"
Postoperative Pain score | 6 hours
  The intensity of pain is evaluated by the visual analog scale (VAS) that measures pain severity expressed on a numerical scale of 0-10: 0, "no pain"; 10, "worst pain imaginable"
Postoperative Pain score | 12 hours
  The intensity of pain is evaluated by the visual analog scale (VAS) that measures pain severity expressed on a numerical scale of 0-10: 0, "no pain"; 10, "worst pain imaginable"
Postoperative Pain score | 24 hours
  The intensity of pain is evaluated by the visual analog scale (VAS) that measures pain severity expressed on a numerical scale of 0-10: 0, "no pain"; 10, "worst pain imaginable"

SECONDARY OUTCOMES:
Additional opioid-type drugs | 24 hours
  The presence of additional opioid analgesic requirements will be evaluated. All patients will be prescribed intravenous analgesia on a strict schedule as follows: ketorolac 30mg in intravenous infusion every 8 hours.
  If the follow-up assessment of postoperative pain is greater than or equal to 4 in the VAS, additional medication is indicated, which is considered as analgesic rescue and which consists of buprenorphine at a dose of 2 mcg kg corrected with 30% according to ideal weight intravenously in both groups, with a dose no greater than 6 mcg / kg / day.
Postoperative nausea and vomiting | 24 hours
  Incidence of postoperative nausea and vomiting (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Jose Camilo Muñoz Chaves, Matamoros, Tamaulipas, Mexico